CLINICAL TRIAL: NCT01671462
Title: European Clinical Evaluation of the BD HPV Assay on the BD Viper LT System
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MDX-11-EUHPV
Record Dates: First submitted 2012-07-13; First posted 2012-08-23 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Uterine Cervical Neoplasms
Keywords: HPV; Cervical Cancer; Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BD HPV assay on Viper LT

SUMMARY:
The purpose of the study is to compare the results of the Becton Dickinson (BD) Human Papilloma Virus (HPV) Assay on the Viper LT instrument from SurePath media diluted in HPV diluent (pre-quot and/or residual), PreservCyt media diluted in HPV diluent (pre-quot and/or residual) and a BD cervical brush in BD transport medium to reference histology results from biopsy.

DETAILED DESCRIPTION:
This is a multicenter study consisting of 2-3 European clinical trial sites, and up to 2 BD Viper LT Systems.

The BD HPV Diluent tube will be run on the BD HPV assay with the Viper LT instrument and compared to histology, Digene hybrid capture 2 (HC2), and Roche LINEAR ARRAY HPV Genotyping Test results.

ELIGIBILITY:
Inclusion Criteria:

* Referred to follow up due to one or more abnormal Pap or an HPV infection
* Subjects who have provided informed consent
* Subjects who meet the minimum age set forth by the ethics committee (EC) and/or national screening guidelines.

Exclusion Criteria:

* Known to be pregnant
* With prior complete or partial hysterectomy involving removal of cervix
* Subjects with an application of chemical compounds to the cervical area 24 hour prior to study entry- this includes acetic acid, iodine, spermicide, douche, anti-fungal meds.
* Subjects on who conization, Loop electrosurgical excision procedure (LEEP), laser surgery or cryosurgery has been performed.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes retrospectively (residual, frozen) collected SurePath or PreservCyt vials and prospectively collected BD cervical brushes in BD transport medium, and SurePath or PreservCyt vials from subjects who meet the inclusion criteria below.
Sampling Method: Non-Probability Sample
Enrollment: 1365 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the BD HPV Assay with 95% confidence intervals for detecting cervical disease as defined by Cervical Intraepithelial Neoplasia (CIN2) or higher. | Nine months
  Sensitivity is calculated: Number of subjects with positive BD HPV test and with histology results of CIN2 or greater divided by the total number of subjects with histology results of CIN2 or greater
Specificity of the BD HPV Assay with 95% confidence intervals for detecting cervical disease as defined by Cervical Intraepithelial Neoplasia (CIN2) or higher. | Nine months
  Specificity is calculated: Number of subjects with a negative BD HPV test and with histology results of less than CIN2 divided by the total number of subjects with histology results of less than CIN2.
Positive Predictive Value (PPV) of the BD HPV Assay with 95% confidence intervals for detecting cervical disease as defined by Cervical Intraepithelial Neoplasia (CIN2) or higher. | Nine months
  Positive Predictive Value is calculated: Number of subjects with a positive BD HPV test and with histology results of CIN2 or greater divided by the total number of subjects with a positive BD HPV test.
Negative Predictive Value (NPV) of the BD HPV Assay with 95% confidence intervals for detecting cervical disease as defined by Cervical Intraepithelial Neoplasia (CIN2) or higher. | Nine months
  Negative Predictive Value is calculated: Number of subjects with a negative result for the BD HPV test and histology results less than CIN2 divided by the total number of subjects with negative results for the BD HPV test.

SECONDARY OUTCOMES:
The positive percent agreement of the BD HPV Assay compared to digene hybrid capture (HC2) test and Roche LINEAR ARRAY HPV Genotyping Test | 9 months
  Positive percent agreement is calculated: The number of subjects with positive BD HPV test and positive results for the HC2 test and Roche Linear Array HPV divided by total of subjects with positive results for HC2 test and Roche Linear Array HPV.
Negative percent agreement of the BD HPV Assay compared to digene hybrid capture (HC2) test and Roche LINEAR ARRAY HPV Genotyping Test | Nine months
  Negative percent agreement is calculated: The number of subjects with negative BD HPV test and negative results for the HC2 test and Roche Linear Array HPV divided by total of subjects with negative results for HC2 test and Roche Linear Array HPV test.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hannet, MD, Study Director — Becton, Dickinson and Company
Locations (2):
- Hvidovre Hospital, Hvidovre, Denmark
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Ejegod DM, Junge J, Franzmann M, Kirschner B, Bottari F, Sideri M, Sandri MT, Bonde J. Clinical and analytical performance of the BD Onclarity HPV assay for detection of CIN2+ lesions on SurePath samples. Papillomavirus Res. 2016 Dec;2:31-37. doi: 10.1016/j.pvr.2016.01.003. Epub 2016 Mar 2. PMID 29074183
- [Derived] Ejegod DM, Rebolj M, Bonde J. Comparison of analytical and clinical performance of CLART HPV2 genotyping assay to Linear Array and Hybrid Capture 2: a split-sample study. BMC Cancer. 2015 Apr 2;15:216. doi: 10.1186/s12885-015-1223-z. PMID 25886410